CLINICAL TRIAL: NCT06681779
Title: A Prospective, Two-phase, Dose-response and Efficacy Study of Transcutaneous Electrical Stimulation As a Noxious Stimulus for the Glasgow Coma Scale
Brief Title: A Study of Transcutaneous Electrical Stimulation As a Noxious Stimulus for the Glasgow Coma Scale
Acronym: GCS02
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Markey Olson (Other)
Responsible Party: Sponsor-Investigator, Markey Olson, Program Manager, St. Joseph's Hospital and Medical Center, Phoenix
Organization: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: 24-500-265-30-06
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Comatose
Keywords: Glasgow Coma Scale; Coma; Transcutaneous stimulation
MeSH Terms: conditions — Coma | interventions — Transcutaneous Electric Nerve Stimulation; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (10):
- E2 (Experimental): Patients with a stable GCS subscore of E2, eyes opening to pain
  Interventions: Device: Transcutaneous electrical stimulation; Other: Standard of Care (SOC)
- E1 (Experimental): Patients with a stable GCS subscore of E2, eyes non-responsive to pain
  Interventions: Device: Transcutaneous electrical stimulation; Other: Standard of Care (SOC)
- Upper Extremity M5 (Experimental): Patients with a stable GCS subscore of M5, localizing, in at least one upper limb
  Interventions: Device: Transcutaneous electrical stimulation; Other: Standard of Care (SOC)
- Upper Extremity M4 (Experimental): Patients with a stable GCS subscore of M4, withdrawing, in at least one upper limb
  Interventions: Device: Transcutaneous electrical stimulation; Other: Standard of Care (SOC)
- Upper Extremity M3 (Experimental): Patients with a stable GCS subscore of M3, flexing, in at least one upper limb
  Interventions: Device: Transcutaneous electrical stimulation; Other: Standard of Care (SOC)
- Upper Extremity M2 (Experimental): Patients with a stable GCS subscore of M2, extending, in at least one upper limb
  Interventions: Device: Transcutaneous electrical stimulation; Other: Standard of Care (SOC)
- Upper Extremity M1 (Experimental): Patients with a stable GCS subscore of M1, no response to stimuli, in at least one upper limb
  Interventions: Device: Transcutaneous electrical stimulation; Other: Standard of Care (SOC)
- Lower Extremity M4 (Experimental): Patients with a stable GCS subscore of M4, withdrawing, in at least one lower limb
  Interventions: Device: Transcutaneous electrical stimulation; Other: Standard of Care (SOC)
- Lower Extremity M3 (Experimental): Patients with a stable GCS subscore of M3, flexing, in at least one lower limb
  Interventions: Device: Transcutaneous electrical stimulation; Other: Standard of Care (SOC)
- Lower Extremity M1 (Experimental): Patients with a stable GCS subscore of M1, no response, in at least one lower limb
  Interventions: Device: Transcutaneous electrical stimulation; Other: Standard of Care (SOC)

INTERVENTIONS:
Device: Transcutaneous electrical stimulation — Transcutaneous electrical stimulation will be used to create noxious stimuli for the GCS exam
Other: Standard of Care (SOC) — Physical pain stimulation, as used in traditional standard care, will be used to score the GCS exam, and the device results will be compared to this SOC exam.

SUMMARY:
The purpose of this study is to determine whether electrical stimulation can be used to replace physical stimulation to test awareness of patients with impaired consciousness. Physical stimulation can cause bruising, damaged nails and ribs, and other damage with repeated testing, and electrical stimulation may be safer and cause less distress with time. This device has not been approved by the U.S. Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
For patients enrolled in this study, the study doctor or study staff will give non-invasive electrical stimulation to measure response. Depending on what study group, the study team may apply this stimulation several times at one (Phase 1) or two (Phase 2) separate time points approximately 2 hours apart (when GCS would normally be collected as part of clinical care). In addition to GCS using normal physical stimulation, the study team will test responses to electrical stimulation. To do this, electrodes (special wired stickers that conduct electricity) will be placed on the forehead, finger, and toe. Stimulation will be applied to one area at a time by connecting the electrode to a stimulator. For each physical and electrical stimulation, response will be measured (such as flinching, opening eyes, making sounds, etc.). The goal is to create electrical stimulation patterns that cause the same response as the physical exam without causing any physical damage.

A video recording will also be taken of the participant's telemetry unit (the screen showing their heart rate and other vital signs throughout the study. This video, in addition to the information from the participant's medical record, is to make sure that there are no unexpected changes in vital signs during the study. The participant will not be visible on this video.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is admitted to the Barrow Neurological Institute's neuro ICU
2. Patient is in a comatose state, which is defined as a patient who is both non-responsive and has a GCS eye or motor response sub-score that requires noxious stimulation
3. Age greater than or equal to 18 years
4. Patient has an available surrogate decision maker with the capacity to consent for participation in a research study

Exclusion Criteria:

1. A neurologic decline immediately prior to study participation that requires urgent or emergent workup or management*
2. Patients in whom the frequency or extent of neurologic assessments is being limited due to concern that noxious stimulation may provoke intracranial hypertension, cardiorespiratory instability, or other adverse events
3. Patients with an implantable or external pacemaker that is currently in use
4. Ongoing refractory cardiorespiratory instability
5. Pregnant females
6. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of Transcutaneous Stimulation Glascow Coma Scale (Exams) score with traditional SOC | Less than 24 hours
  Two GCS exams will be conducted at the same time point, and it will be determined whether the same score is obtained for both methods.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon M Fox, MD, PhD, Study Director — Barrow Neurological Institute
Locations (1):
- Barrow Neurological Institute, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No